CLINICAL TRIAL: NCT00782236
Title: Comparison of an Alloplast (Straumann Bone Ceramic) to an Allograft of Freeze Dried Bone (FDBA) for Preservation of the Alveolar Ridge Following Tooth Extraction: a Prospective, Randomized, Controlled Clinical Study
Brief Title: Comparison of Straumann BoneCeramic vs. Allograft Bone in Extraction Sockets
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Institut Straumann AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR 02/06
Record Dates: First submitted 2008-10-28; First posted 2008-10-31 (Estimated); Last update posted 2016-03-04 (Estimated); Status verified 2016-03

CONDITIONS: Tooth Loss
MeSH Terms: conditions — Tooth Loss | interventions — Bone Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Straumann BoneCeramic (Active Comparator): In the test group, the subjects will receive the Bone Graft Material Straumann BoneCeramic in combination with a collagen membrane for preservation of the alveolar ridge after tooth extraction.
  Interventions: Device: Bone Graft Material
- Freeze Dried Allograft Bone (Active Comparator): In the control group, the subjects will receive Bone Graft Material Freeze Dried Allograft Bone in combination with a collagen membrane for preservation of the alveolar ridge after tooth extraction.
  Interventions: Device: Bone Graft Material

INTERVENTIONS:
Device: Bone Graft Material — After screening and enrollment, subjects will undergo tooth extraction of a single tooth with placement of Straumann Bone Ceramic or Freeze Dried Allograft Bone (FDBA) with a resorbable collagen membrane (Bio-Gide) for preservation of the alveolar ridge following tooth extraction. Following 6 months of healing, a core of bone will be taken from the surgical site and a dental implant will be placed. The subjects will then be followed for 12 months following dental implant placement.
  Other Names: Synthetic bone substitute; Allograft bone

SUMMARY:
The primary objective of this study is to evaluate the implant stability at the time of abutment placement on implants placed in healed extraction sockets treated with Straumann BoneCeramic (SBC) versus Freeze Dried Bone Allograft (FDBA).

DETAILED DESCRIPTION:
Subjects will undergo a single tooth extraction and then will be randomized to receive SBC or FDBA. Following a healing period of 6 months, a core biopsy will be taken of the augmented site and a dental implant will be placed. The subject will be followed for one year following dental implant placement for implant success and survival.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have voluntarily signed the informed consent form
* Subjects must be between the ages of 18 and 80
* Subjects must need a single tooth extraction in ADA sites 3-6 and 11-14 without septal bone in the maxilla and in ADA sites 19-30 without septal bone in the mandible and would benefit from prosthetic reconstruction with a dental implant
* Subjects must be committed to the study and the required follow-up visits
* Subjects must be in good general health as assessed by the Investigator

Exclusion Criteria:

* Presence of conditions requiring chronic routine prophylactic use of antibiotics
* Pregnancy
* Medical conditions requiring prolonged use of steroids
* History of leukocyte dysfunction and deficiencies
* History of bleeding disorders
* History of neoplastic disease requiring the use of chemotherapy
* History of radiation therapy to the head and neck
* Subjects with a history of renal failure
* Subjects with severe or uncontrolled metabolic bone disorders
* Uncontrolled endocrine disorders
* Subjects who knowingly have HIV or hepatitis
* Physical handicaps that would interfere with the ability to perform adequate oral hygiene
* Subjects who have undergone administration of any investigational drug or device within 30 days of enrollment in the study
* Alcoholism or drug abuse
* Subjects who are heavy smokers (>10 cigarettes per day or cigar equivalents) or chew tobacco
* Conditions or circumstances, in the opinion of the Investigator, which would prevent completion of study participation or interfere with analysis of study results, such as history of non-compliance or unreliability
* Local inflammation including untreated periodontitis
* Mucosal diseases such as erosive lichen planus
* History of local radiation therapy
* Presence of oral lesions (such as ulcerations or malignancy)
* Bone defects that exclude implant restoration
* Subjects who have a full mouth plaque level >30% at the baseline visit
* Severe bruxing or clenching habits
* Persistent intra-oral infection
* Subjects presenting with an acute abscess in the tooth to be extracted or in the adjacent teeth to the extraction site (sites with presence of asymptomatic chronic lesions are eligible)
* Subjects with inadequate oral hygiene or unmotivated for adequate home care
* At the time of tooth extraction, if any bony wall is severely damaged or completely lost (i.e., anything other than a four wall extraction socket)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2006-06; Primary Completion 2007-11 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Implant stability will be assessed by recording the maximum torque achieved when placing the abutment. The implant will be considered stable if a minimum of 35 Ncm of torque is achieved. | Six weeks following dental implant placement

SECONDARY OUTCOMES:
Histological evaluation | 6 months following tooth extraction
Alveolar ridge width and height changes | 6 months following tooth extraction
Periodontal measurements | 6 months following tooth extraction and 6 and 12 months following implant placement
Grafting procedure success rate | 14 days, 1 month, 3 months, and 6 months following tooth extraction
Implant success and survival rate | 6 weeks, 12 weeks, 6 months, and 12 months following implant placement
Mesial and distal implant bone level changes | 6 weeks, 12 weeks, 6 months, and 12 months following implant placement
Patient satisfaction | 6 and 12 months following implant placement

CONTACTS AND LOCATIONS:
Overall Officials: Paul S. Rosen, DMD, MS, Principal Investigator — Private Practice
Locations (1):
- Private Practice, Yardley, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No